CLINICAL TRIAL: NCT03512899
Title: Internal Jugular Vein Versus Axillary Vein With Single-incision for Implantable Ports: a Prospective and Randomized Study.
Brief Title: Comparison Between Internal Jugular Vein Versus Axillary Vein for Implantable Ports
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AC Camargo Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 63850017.5.0000.5432
Record Dates: First submitted 2018-02-06; First posted 2018-05-01 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2021-01

CONDITIONS: Catheter Complications; Cancer
Keywords: implantable port
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Comparison between internal jugular vein versus via axillary vein with single-incision for placement of implantable ports in cancer patients. Investigators are recruiting 240 patients and randomizing 120 for each arm. Primary outcome is early complications, until 30 days and secondary outcome late complications, between 30 days and 6 months. The follow-up is 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal jugular vein access (Active Comparator): Internal jugular vein access preferably right, assisted by ultrasound and radioscopy. Catheter: districath®, 8.5 French.
  Interventions: Procedure: Right internal jugular access.; Procedure: Left internal jugular access.
- Axillary vein access (Active Comparator): Axillary vein access with single incision, assisted by ultrasound and radioscopy. Catheter: districath®, 8.5 French.
  Interventions: Procedure: Right axillary vein access.; Procedure: Left axillary vein access.

INTERVENTIONS:
Procedure: Right internal jugular access. — Implantation using percutaneous puncture.
  Arms: Internal jugular vein access
Procedure: Left internal jugular access. — Implantation using percutaneous puncture.
  Arms: Internal jugular vein access
Procedure: Right axillary vein access. — Implantation using percutaneous puncture.
  Arms: Axillary vein access
Procedure: Left axillary vein access. — Implantation using percutaneous puncture.
  Arms: Axillary vein access

SUMMARY:
Comparison between internal jugular vein versus via axillary vein with single-incision for placement of implantable ports in cancer patients. Investigators are recruiting 240 patients and randomizing 120 for each arm. Primary outcome is early complications, until 30 days and secondary outcome late complications, between 30 days and 6 months. The follow-up is 12 months.

DETAILED DESCRIPTION:
Prospective and randomized trial comparing internal jugular vein versus via axillary vein with single-incision for placement of implantable ports in cancer patients. Investigators are recruiting 240 patients and randomizing 120 for each arm in a single center study at AC Camargo Cancer Center. Every surgery is assisted by ultrasound and radioscopic and the catheter is districath®, 8.5 French. Clinical assessment will be at 10 days and every 3 months after surgery. Primary outcome is early complications, until 30 days and secondary outcome late complications, between 30 days and 6 months. The follow-up is 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Catheter due to chemotherapy.
* Cancer patients.
* ECOG (performance status) from 0 to 2.
* Signed informed consent form.

Exclusion Criteria:

* Non compliance.
* Anticoagulant therapy.
* Coagulopathy (platelet count below 50,000 and/or protrombin time above 18s).
* Death within 30 days after the procedure.
* Another catheter in superior vena cava.
* Previous long term catheter in superior vena cava.
* Obesity (IBM>40 Kg/m2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Early complications. | 30 days
  Early complications within 30 days during clinical assessment. These outcomes are divided in intra-operative complications, such as pneumothorax, hemothorax, vascular injury, cardiac arrhythmia, hematoma; and post-operative until 30 days complications such as wound infections, catheter related bacteremia, catheter disfunction, catheter related deep venous thrombosis, reservoir extrusion and skin erosion.

SECONDARY OUTCOMES:
Late complications | 30 to 180 days
  Post-operative between 30 days and 6 months complications such as wound infections, catheter related bacteremia, catheter disfunction, catheter related deep venous thrombosis, reservoir extrusion and skin erosion.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno S Pignataro, Principal Investigator — Vascular and Endovascular Surgery Department
Locations (1):
- AC Camargo Cancer Center, São Paulo, Brazil